CLINICAL TRIAL: NCT02963389
Title: A Phase I Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Tripegfilgrastim After Single Administration in Pediatric Solid Tumor/Lymphoma Patients
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Tripegfilgrastim in Pediatric Solid Tumor/Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA3031_PNP_I
Record Dates: First submitted 2016-10-13; First posted 2016-11-15 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor, human

ARMS (4):
- Tripegfilgrastim 60ug/kg, >=6 and <12-year-old patients (Experimental): A single dose of Tripegfilgrastim 60ug/kg, S.C, 24hr after completion of chemotherapy
  Interventions: Drug: Tripegfilgrastim
- Tripegfilgrastim 60ug/kg, >=12 and <19-year-old patients (Experimental): A single dose of Tripegfilgrastim 60ug/kg, S.C, 24hr after completion of chemotherapy
  Interventions: Drug: Tripegfilgrastim
- Tripegfilgrastim 100ug/kg, >=6 and <12-year-old patients (Experimental): A single dose of Tripegfilgrastim 100ug/kg, S.C, 24hr after completion of chemotherapy
  Interventions: Drug: Tripegfilgrastim
- Tripegfilgrastim 100ug/kg, >=12 and <19-year-old patients (Experimental): A single dose of Tripegfilgrastim 100ug/kg, S.C, 24hr after completion of chemotherapy
  Interventions: Drug: Tripegfilgrastim

INTERVENTIONS:
Drug: Tripegfilgrastim
  Other Names: DA-3031

SUMMARY:
This is an open-label, single ascending dose study to evaluate safety, tolerability, and pharmacokinetics/pharmacodynamics of Tripegfilgrastim in pediatric solid tumor/lymphoma patients

ELIGIBILITY:
Inclusion Criteria:

* >=6 and <19-year-old pediatrics with solid tumor/lymphoma
* Scheduled for chemotherapy requiring G-CSF support or having given an experience of ANC < 0.5x10^9/L
* ANC > 0.75x10^9/L, platelet > 75x10^9/L
* ECOG performance status 0 or 1

Exclusion Criteria:

* Patients with leukemia, myelodysplastic syndrome or uncontrolled infectious/nervous diseases
* History of allergy to filgrastim, pegfilgrastim or known hypersensitivity to E-coli derived proteins.
* Women who are pregnant or lactating

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
PK parameter | Day 1(Hour 0) ~ Day 21
  Time to reach Cmax of Tripegfilgrastim [Tmax]
PK parameter | Day 1(Hour 0) ~ Day 21
  Peak plasma concentration of Tripegfilgrastim [Cmax]
PK parameter | Day 1(Hour 0) ~ Day 21
  Area under the plasma concentration of Tripegfilgrastim versus time curve [AUC]
PK parameter | Day 1(Hour 0) ~ Day 21
  Half-life of Tripegfilgrastim [T1/2]
PK parameter | Day 1(Hour 0) ~ Day 21
  The lowest plasma concentration that Tripegfilgrastim reaches before the next dose is administered [Ctrough]

SECONDARY OUTCOMES:
PD parameter | Day 1(Hour 0) ~ Day 14
  Peak plasma concentration of Absolute Neutrophil Count [ANCmax]
PD parameter | Day 1(Hour 0) ~ Day 14
  Area under the plasma concentration of Absolute Neutrophil Count versus time curve [AUC(ANC)]
PD parameter | Day 1(Hour 0) ~ Day 14
  Time to reach Cmax of Absolute Neutrophil Count [Tmax(ANC)]

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee S, Hong KT, Jang IJ, Yu KS, Kang HJ, Oh J. Semimechanistic pharmacokinetic-pharmacodynamic model of tripegfilgrastim for pediatric patients after chemotherapy. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1319-1334. doi: 10.1002/psp4.13012. Epub 2023 Aug 9. PMID 37559343
- [Derived] Lee S, Hong KT, Moon SJ, Choi JY, Hong CR, Shin HY, Cho JY, Jang IJ, Yu KS, Oh J, Kang HJ. Pharmacokinetic and Pharmacodynamic Characteristics of Tripegfilgrastim, a Pegylated G-CSF, in Pediatric Patients with Solid Tumors. Clin Pharmacol Ther. 2022 Jan;111(1):293-301. doi: 10.1002/cpt.2433. Epub 2021 Oct 27. PMID 34605552